CLINICAL TRIAL: NCT05192122
Title: Free From Maintenance Drug Therapy in Multiple Myeloma (The FREEDMM Trial): A Pilot Study of Minimal Residual Disease (MRD)-Driven Discontinuation of Maintenance (HEME-20)
Brief Title: Free From Maintenance Drug Therapy in Multiple Myeloma (The FREEDMM Trial) for Minimal Residual Disease (MRD
Acronym: HEME-20
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Karen Sweiss, Principal Investigator, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1196
Record Dates: First submitted 2022-01-07; First posted 2022-01-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Patients with sustained MRD negativity (defined as MRD negative at 2 time points, at least 12 months apart) will stop maintenance therapy. Bone marrow MRD testing must be performed at UIC prior to study entry can be counted as the first time point as long as the patient has received at least 2 years of maintenance at the time of MRD testing.
  These patients will then be monitored for sustained MRD-negativity after stopping therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone marrow MRD-negative VGPR or CR (Other): Discontinue maintenance therapy after at least three years
  Interventions: Other: Discontinue maintenance therapy SOC
- Bone marrow MRD-positive VGPR or CR (Other): Continue maintenance therapy as per SOC
  Interventions: Other: Discontinue maintenance therapy SOC

INTERVENTIONS:
Other: Discontinue maintenance therapy SOC — MRD testing through NGS Clonoseq will be performed as standard of care on all bone marrow samples. MRD negativity will be defined as observation of no templates at a sensitivity of 1 in a 1,000,000 (10-6) cells assessed, with a minimum of 1 million cells undergoing assessment. In addition, patients must be in VGPR/CR/PR as defined previously.

SUMMARY:
A pilot study to assess the risk of progression after stopping post-autologous stem cell transplant (ASCT) maintenance therapy in Minimal Residual Disease (MRD)-negative MM patients.

DETAILED DESCRIPTION:
This is a pilot study to assess the risk of progression after stopping post-autologous stem cell transplant (ASCT) maintenance therapy in Minimal Residual Disease (MRD)-negative Multiple Myeloma (MM) patients. Patients will be eligible if they have a diagnosis of active MM, have completed at least 2 years of maintenance therapy post-ASCT, and meet International Myeloma Working Group (IMWG) criteria for very good partial response (VGPR) or complete response (CR). Once eligibility is confirmed and informed consent is signed, MRD testing will be performed on routine bone marrow aspirate using standard of care next-generation sequencing (NGS) testing and will be defined at a threshold of 10-6. Patients who are in VGPR or CR and sustained MRD (defined as MRD-negative at two time points that are at least 1 year apart) will go on to discontinue maintenance therapy. MRD-positive patients will continue to be treated as per standard of care (i.e., continue maintenance). Both MRD-positive and MRD-negative patients will be followed as per standard of care for progression using IMWG criteria and for MRD. Quality of life will be assessed at baseline and at 3 months after discontinuing maintenance therapy in MRD-negative patients and at baseline and at the time of next follow-up after MRD testing in MRD-positive patients. In patients who stop maintenance therapy, MRD status will be re-assessed by yearly bone marrow aspirate as per standard of care. Treatment for relapsed/ refractory myeloma will be instituted at the treating physician's discretion for documented clinical and/or biochemical progression. For all patients, a 5-mL peripheral blood and bone marrow sample will be collected and stored at the time of each standard of care bone marrow biopsy and at time of documented disease progression for correlative testing.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status equal to or less than 2 within 30 days prior to registration
* Revised International Staging System (R-ISS) I,2 or 3
* Patients with multiple myeloma as defined by IMWG
* Received at least 2 years of post ASCT maintenance (patients may have received any number of prior lines of therapy).
* Maintenance therapy is defined as any anti-myeloma therapy initiated after ASCT to prevent disease recurrence and prolong time in remission (i.e., lenalidomide, bortezomib, RVD, etc.)
* Disease response is VGPR or CR at the time of enrollment as defined by IMWG criteria.
* Patients or their legally authorized representative must be able to understand and be willing to sign a voluntary informed consent form and agree to compliance with the protocol schedule; with the knowledge that they may withdraw consent at any time without impact on future medical care

Exclusion Criteria:

* Patients with plasma cell leukemia, AL amyloidosis or Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, Skin (POEMS) syndrome
* Prior organ transplant or condition requiring immunosuppressive therapy
* Prior allogeneic hematopoietic cell transplant
* Treatment with any investigational drug within 30 days prior to enrollment
* Unable to sign an informed consent or their legally authorized represnetative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have a sustained MRD-negative VGPR or CR measured by a bone marrow biopsy | 12 months after stopping maintenance therapy
  Number of participants that have a sustained MRD-negative VGPR or CR measured by a bone marrow biopsy (MRD defined as 10-6)

SECONDARY OUTCOMES:
Number of participants that have a sustained MRD-negative VGPR or CR measured by a bone marrow biopsy | 2 years after stopping maintenance therapy
  Number of participants that have a sustained MRD-negative VGPR or CR measured by a bone marrow biopsy (MRD defined as 10-6)
Number of participants that relapse per IMWG at 1 year after stopping maintenance therapy | 1 year after stopping maintenance therapy
  Number of participants that relapse per IMWG
Number of participants that relapse per IMWG at 2 years after stopping maintenance therapy | 2 years after stopping maintenance therapy
  Number of participants that relapse per IMWG
Progression-free survival (PFS) in multiple myeloma patients | I year
  PFS in multiple myeloma patients at 1 year
Progression-free survival (PFS) in multiple myeloma patients | 2 years
  PFS in multiple myeloma patients at 2 years
Progression-free survival (PFS) in multiple myeloma patients | 3 years
  PFS in multiple myeloma patients at 3 years
Compare health-related quality of life (HRQoL) between MM patients stopping versus continuing maintenance therapy | Baseline
  Compare health-related quality of life (HRQoL) between MM patients stopping versus continuing maintenance therapy therapy using the European Organization for Research and Treatment of Cancer Quality of Life Multiple Myeloma questionnaire (EORTC QLQ-MY20) questionnaire
Compare health-related quality of life (HRQoL) between MM patients stopping versus continuing maintenance therapy | 3 months
  Compare health-related quality of life (HRQoL) between MM patients stopping versus continuing maintenance therapy using the European Organization for Research and Treatment of Cancer Quality of Life Multiple Myeloma questionnaire (EORTC QLQ-MY20) questionnaire
Correlate peripheral blood circulating myeloma cell numbers (CELLSEARCH) with conventional IMWG response | 1 year
  Measuring the disease response
Correlate peripheral blood circulating myeloma cell numbers (CELLSEARCH) with conventional IMWG response | 2 years
  Measuring the disease response
Correlate peripheral blood circulating myeloma cell numbers (CELLSEARCH) with conventional IMWG response | 3 years
  Measuring the disease response
Correlate peripheral blood circulating myeloma cell numbers (CELLSEARCH) with conventional IMWG response | 1 year
  PFS in multiple myeloma patients at 1 year
Correlate peripheral blood circulating myeloma cell numbers (CELLSEARCH) with conventional IMWG response | 2 years
  PFS in multiple myeloma patients at 2 years
Correlate peripheral blood circulating myeloma cell numbers (CELLSEARCH) with conventional IMWG response | 3 years
  PFS in multiple myeloma patients at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sweiss, PhamD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States